CLINICAL TRIAL: NCT04572945
Title: Foot Abnormalities in Diabetic Patients With and Without Chronic Kidney Disease in Assuit University Hospitals; Case Control Study
Brief Title: Foot Abnormalities in Diabetic CKD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Usra Mohamed Farrag Ahmed, Principal Investigator, Assiut University
Other Study IDs: Diabetic Foot in CKD patients
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: CKD; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Kidney Function Tests; Urinalysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1- Cases: Diabetic patients with CKD.: classified according to estimated GFR into 5 stages according to KIDGO 2012 classification.
  Interventions: Diagnostic Test: kidney function test
- 2- Controls: Diabetic patients without CKD.: defined as patients who have normal kidney function test, normal urine analysis and normal ultrasound findings.
  Interventions: Diagnostic Test: kidney function test

INTERVENTIONS:
Diagnostic Test: kidney function test — laboratory and imaging
  Other Names: HB A1c; urine analysis; abd us

SUMMARY:
1. To find the correlation between different stages of CKD and type and severity of foot abnormalities in diabetic patients with CKD.
2. To assess factors that may aggravate foot abnormalities in diabetic patients with CKD by measuring serum calcium, phosphorus, parathyroid hormone, albumin, uric acid…etc.

DETAILED DESCRIPTION:
Chronic kidney disease is an important contributor to morbidity and mortality, the global prevalence of CKD was 9.1% (697.5 million cases) in 2017(1). Diabetes is a leading cause of end stage renal disease worldwide. (2) Foot abnormalities and amputation are major health concerns as they diminish health-related quality of life and cause financial burden (3).

KDIGO 2020 defines Chronic Kidney Disease (CKD) as persistently elevated urine albumin excretion (≥30 mg/g [3mg/mmol] creatinine), persistently reduced estimated glomerular filtration rate (eGFR <60 ml/min per 1.73 m2), or both, for greater than 3 months. (4) Diabetic foot is defined as either diabetic peripheral neuropathy, peripheral arterial disease, infection, ulceration, or Charcot osteoarthropathy, or a combination of these abnormalities, in a person diagnosed with diabetes mellitus, according to the guidelines of International Working Group of Diabetic Foot 2020 (IWGDF). (5) There is a much higher incidence of diabetic foot disorder in those with renal disease and outcomes are generally poorer (2) as CKD patients are sharing three main risk factors of foot ulceration and amputation: neuropathy, peripheral arterial disease and increased susceptibility to infection with impaired wound healing. (6)

this research is conducted as little is known about the potential relationship between chronic kidney disease and diabetic foot. This research evaluates the true burden of different diabetic foot lesions in CKD patients, assesses the severity of diabetic foot in different stages of CKD and the factors that may aggravate it in CKD, for future need to modify our clinical policies in management of diabetic foot in CKD patients to provide better prognosis and prevent long term disabilities.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic CKD patients classified according to estimated GFR into 5 stages according to KIDGO 2012 classification:

   Stage 1 CKD: eGFR 90 or Greater Stage 2 CKD: eGFR Between 60 and 89 Stage 3 CKD: eGFR Between 30 and 59 Stage 4 CKD: eGFR Between 15 and 29 Stage 5 CKD: eGFR Less than 15 etheir on dialysis ( satge 5 D) or not (stage 5 non D)
2. Age more than ≥18 years

Exclusion Criteria:

1. Patients administer drugs causing neuropathy as:amiodarone, chemotherapy, oxazolidinone linezolid, isoniazid, metronidazole, nitrofurantoin ,immunosuppressants, nucleoside reverse transcriptase inhibitors, levodopa and antifungal drugs.
2. Patients with other causes of CKD.
3. Patients have other causes of PVD.
4. Age less than ˂18 years.
5. Patients' refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * The research includes patients recruited from Internal Medicine department Assiut University Hospitals( renal and dialysis unit and diabetes and endocrinal center) , classified into two groups :
    1. diabetic CKD patient (stage 1- stage 5 non D )
    2. diabetic CKD patient (stage 5 D)
  * written or verbal consent should be taken from those patients that participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of foot abnormalities in diabetic CKD patient | 1 year
  Percentage of foot abnormalities in diabetic CKD patient in different stages according to KIDGO 2012 classification

CONTACTS AND LOCATIONS:
Overall Officials: usra mo farrag, M.B.B.ch, Principal Investigator — eygpt

REFERENCES:
- [Background] Carney EF. The impact of chronic kidney disease on global health. Nat Rev Nephrol. 2020 May;16(5):251. doi: 10.1038/s41581-020-0268-7. No abstract available. PMID 32144399
- [Background] Valabhji J. Foot problems in patients with diabetes and chronic kidney disease. J Ren Care. 2012 Feb;38 Suppl 1:99-108. doi: 10.1111/j.1755-6686.2012.00284.x. PMID 22348369
- [Background] Ndip A, Lavery LA, Boulton AJ. Diabetic foot disease in people with advanced nephropathy and those on renal dialysis. Curr Diab Rep. 2010 Aug;10(4):283-90. doi: 10.1007/s11892-010-0128-0. PMID 20532700
- [Background] Hammond N, Wang Y, Dimachkie MM, Barohn RJ. Nutritional neuropathies. Neurol Clin. 2013 May;31(2):477-89. doi: 10.1016/j.ncl.2013.02.002. PMID 23642720